CLINICAL TRIAL: NCT03124797
Title: Accuracy of SpO2 for Noninvasive Pulse Oximeter Sensor (RD DCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR30835-123A-123B-127A
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RD DCI Sensor (Experimental): All subjects are enrolled into the test group and all subjects received the RD DCI Sensor
  Interventions: Device: RD DCI Sensor

INTERVENTIONS:
Device: RD DCI Sensor — Noninvasive pulse oximeter sensor

SUMMARY:
In this study, the level of oxygen within the blood will be reduced in a controlled manner by reducing the concentration of oxygen the study volunteer breathes. The accuracy of a noninvasive pulse oximeter sensor will be assessed by comparison to the oxygen saturation measurements from a laboratory blood gas analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Competent non-smoking adults between the ages of 18 and 45 for each series of tests.
* Must weigh a minimum of 110 pounds and no more than 250 pounds unless subject is over 6 feet tall.
* Subjects must understand and consent to be in the study.
* American Society of Anesthesiology Class 1 (Healthy subjects without any systemic disease at all).
* Subjects with hemoglobin greater than or equal to 11 g/dL.

Exclusion Criteria:

* Subjects with polished, gel or acrylic nails.
* Subjects with damaged and/or finger nail deformities.
* Subjects who have had caffeine consumption the day of the study.
* Subjects who have taken pain medication 24 hours before the study.
* Subjects who have any systemic disease at all.
* Subjects who do not understand the study and the risks.
* Subjects who smoke.
* Subjects who use recreational drugs.
* Subjects who are pregnant or nursing.
* Subjects having either signs or history of peripheral ischemia.
* Subjects with open wounds, lacerations, inflamed tattoos or piercings, visible healing wounds.
* Subjects with psychiatric conditions or are on psychiatric medications.
* Subjects who have had invasive surgery within the past year- including but not limited to major dental surgery, gallbladder, heart, appendix, major fracture repairs (involving plates/ screws), jaw surgery, Urinary tract surgery, plastic surgery, major ENT surgery, joint replacement or gynecological surgeries.
* Subjects who have had minor surgery or conditions in the past two months including but not limited to minor foot surgery (bunion), arthroscopic procedure, blood donation, plasma donation, skin biopsy/ procedures, root canal, fractures, eye surgery, and other minor procedures.
* Subjects that have been on antibiotics had congestion, head colds, flu, ear infection, chest congestion will have a 2 week waiting period from the time of finishing medications or must have no more symptoms.
* Subjects with claustrophobia, or anxiety.
* Subjects who have been in severe car accidents or a similar type of accidents will have a 12 month waiting period, from the time of the accident.
* Subjects who have had a concussion will have a 12 month waiting period, from the time of the concussion.
* Subjects with chronic unresolved asthma, lung disease and respiratory disease.
* Allergies to lidocaine, latex, adhesives, or plastic.
* Subjects with finger deformities or injuries (specific finger will not be used).
* Subjects with heart conditions, diabetes or hypertension.
* Subjects with resting heart rates greater than 85BPM or below 45BPM
* Subjects who have given birth naturally will have 6 month waiting period. Subjects who had a pregnancy terminated, a miscarriage or had a c-section will have a 12 month waiting period.
* Others deemed ineligible by the clinical staff.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-02; Primary Completion 2016-04-05 (Actual); Study Completion 2016-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RD DCI Sensor
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RD DCI Sensor
Number analyzed (Participants) | 18
Age, Customized [Count of Participants; unit: Participants]
  22-43 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Arms Calculation
Description: Accuracy will be determined by comparing the noninvasive blood oxygen saturation measurement of the pulse oximeter to that obtained from a blood sample and calculating the arithmetic root mean square(Arms) error value. In order to obtain the Arms value, the blood oxygen saturation measurement is subtracted from the pulse oximeter oxygen saturation measurement for a number of samples, the average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: 1-5 hours
Measure: Number; unit: % of oxygen saturated hemoglobin
Units Other Than Participants: data points
Arm/Group | RD DCI Sensor
Number analyzed (Participants) | 18
Number analyzed (data points) | 492
% of oxygen saturated hemoglobin | 1.9

ADVERSE EVENTS:
Arm/Group | RD DCI Sensor
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RD DCI Sensor (N=18)
Arterial line site sensitivity (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes